CLINICAL TRIAL: NCT00470665
Title: An Open-Label, Concentration-Controlled, Randomized, 12-Month Study of Prograf + Rapamune + Corticosteroids Compared to Cyclosporine,USP (Modified) + Rapamune + Corticosteroids in High Risk Renal Allograft Recipients
Brief Title: Study Comparing Sirolimus/Prograf vs Sirolimus/CsA in High-Risk Renal Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0468H1-903
Record Dates: First submitted 2007-05-07; First posted 2007-05-08 (Estimated); Last update posted 2007-05-08 (Estimated); Status verified 2007-05

CONDITIONS: Renal Allograft Recipients
MeSH Terms: interventions — Sirolimus

INTERVENTIONS:
Drug: Rapamune

SUMMARY:
The purpose of this study is to assess whether in high-risk kidney transplant patients (patients whose previous kidney transplant failed, have a high PRA lab test result or are of African-American descent) that a combination of Rapamune with Prograf and steroids will prevent acute rejection as well as Rapamune and cyclosporine and steroids.

ELIGIBILITY:
Inclusion criteria:

* Patients of African-American descent or patient with a history of multiple transplants and/or patients with a high panel reactive antibody lab test with a renal transplant from a cadaveric donor, a living unrelated donor or a living-related mismatched donor.
* Age >= 13 years, weight >= 40 kg
* Women must have a negative pregnancy test at study entry

Exclusion criteria

* Multiple organ transplants or double kidney transplants (pediatric en-bloc or double adult)
* Active systemic infection, or localized major infection or known HIV
* Patients with residual kidney function >20 mL/min

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 460
Dates: Start 2002-08; Study Completion 2004-07

PRIMARY OUTCOMES:
First biopsy-confirmed acute rejection, patient death or graft loss in the first 12 months following transplantation. First occurence of kidney graft loss or patient death in the first 12 months following transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Oliveras L, Lopez-Vargas P, Melilli E, Codina S, Royuela A, Coloma Lopez A, Fava A, Manonelles A, Couceiro C, Lloberas N, Cruzado JM, Montero N. Delayed initiation or reduced initial dose of calcineurin-inhibitors for kidney transplant recipients at high risk of delayed graft function. Cochrane Database Syst Rev. 2025 Apr 8;4(4):CD014855. doi: 10.1002/14651858.CD014855.pub2. PMID 40197799
- [Derived] Gaber AO, Kahan BD, Van Buren C, Schulman SL, Scarola J, Neylan JF; Sirolimus High-Risk Study Group. Comparison of sirolimus plus tacrolimus versus sirolimus plus cyclosporine in high-risk renal allograft recipients: results from an open-label, randomized trial. Transplantation. 2008 Nov 15;86(9):1187-95. doi: 10.1097/TP.0b013e318187bab0. PMID 19005398